CLINICAL TRIAL: NCT02533674
Title: Phase I Multicenter, Open-label, Clinical and Pharmacokinetic Study of PM060184 in Combination With Gemcitabine in Selected Patients With Advanced Solid Tumors
Brief Title: Multicenter, Open-label, Clinical and Pharmacokinetic Study of PM060184 in Combination With Gemcitabine in Selected Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PharmaMar (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PM60184-A-003-14; PM60184-A-003-14 (Other: Pharma Mar USA, Inc.); 2014-002943-16 (EudraCT Number)
Record Dates: First submitted 2015-08-07; First posted 2015-08-27 (Estimated); Results first posted 2021-05-13 (Actual); Last update posted 2021-06-11 (Actual); Status verified 2021-05

CONDITIONS: Solid Tumors
MeSH Terms: interventions — Gemcitabine; plocabulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- gemcitabine plus PM060184 (Experimental)
  Interventions: Drug: Gemcitabine plus PM060184

INTERVENTIONS:
Drug: Gemcitabine plus PM060184

SUMMARY:
Prospective, open-label, dose-ranging, uncontrolled phase I study with escalating doses of PM060184 in combination with gemcitabine in selected patients with advanced solid tumors.

The study objectives are:

To determine the MTD and the RD of PM060184 in combination with gemcitabine in selected patients with advanced solid tumors.

To characterize the safety profile and feasibility of this combination in this study population.

To characterize the pharmacokinetics of this combination and to detect major drug-drug PK interactions.

To obtain preliminary information on the clinical antitumor activity of this combination.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed and dated written informed consent prior to any specific study procedure.
2. Age ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 1 (see APPENDIX 1).
4. Life expectancy ≥ 3 months.
5. Patients with a histologically/cytologically confirmed diagnosis of advanced disease of any of the following tumors that progressed to standard therapy or for whom no standard therapy exists:

   * Breast cancer non-candidate for hormone therapy alone.
   * Epithelial ovarian cancer (including primary peritoneal disease and/or fallopian tube carcinomas and/or endometrial adenocarcinomas).
   * Locally advanced or metastatic head and neck cancer.
   * Non-small cell lung cancer (NSCLC).
   * Germ cell tumors (GCTs).
   * Biliary tract adenocarcinoma.
   * Adenocarcinoma or carcinoma of unknown primary site (UKPS).
   * Cervix carcinoma.
   * Gastrointestinal stromal tumor (GIST).
   * Urothelial cancer.
6. Expansion cohort at the RD:

   All patients must have:
   * Measurable disease according to RECIST v.1.1 (or Choi criteria and/or EORTC metabolic response criteria for solid tumors, in the case of GIST); or
   * Evaluable disease by serum markers in the case of ovarian cancer [Gynecologic Cancer Intergroup (GCIG) specific criteria]; and
   * Documented disease progression during or immediately after last therapy according to any of the aforementioned criteria.
7. Wash-out periods: at least three weeks since the last anticancer therapy, including radiation therapy (RT) in more than 35% of the bone marrow; at least three weeks since the last biological/investigational therapy [excluding monoclonal antibodies (MAbs)]; at least four weeks since the last MAb-containing therapy; and at least six weeks since nitrosoureas and mitomycin C (systemic). In the case of hormonesensitive breast cancer progressing while on hormone therapy, the latter must be either stopped up to one week before or continued without changes during the trial.
8. Adequate bone marrow, renal, hepatic, and metabolic function (assessed ≤ 7 days before inclusion in the study):

   * Platelet count ≥ 100 x 109/l, hemoglobin ≥ 9.0 g/dl and ANC ≥ 1.0 x 109/l.
   * AST and ALT ≤ 3.0 x ULN, independently of the presence of liver metastases.
   * AP ≤ 2.5 x ULN (≤ 5 x ULN if disease-related).
   * Total bilirubin ≤ 1.5 x ULN.
   * International Normalized Ratio (INR) < 1.5 (except if patient is on oral anticoagulation therapy).
   * Calculated creatinine clearance (CrCl) ≥ 50 ml/minute (using Cockcroft and Gault's formula; see APPENDIX 2).
   * Albumin ≥ 2.5 g/dl.
9. Recovery to grade ≤ 1 from any AE derived from previous treatment (excluding alopecia and/or cutaneous toxicity and/or asthenia).
10. Left ventricular ejection fraction (LVEF) by echocardiography (ECHO) or multiplegated acquisition (MUGA) within normal range (according to institutional standards).
11. Women of childbearing potential must have a negative serum or urine pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for six weeks after discontinuation of treatment. Acceptable methods of contraception include intrauterine device (IUD), oral contraceptive, subdermal implant and/or double barrier.

Exclusion Criteria:

1. Concomitant diseases/conditions:

   * History or presence of unstable angina, myocardial infarction, congestive heart failure, or clinically significant valvular heart disease within last year.
   * Symptomatic arrhythmia or any uncontrolled arrhythmia requiring ongoing treatment.
   * Known chronic active hepatitis or cirrhosis
   * Active uncontrolled infection [i.e., antibiotic, antifungal or antiviral intervention indicated or surgical procedure (i.e., pleural or deep abscess drainage) conducted within 15 days prior to inclusion].
   * Known human immunodeficiency virus (HIV) infection.
   * Current or prior history of grade ≥ 2 peripheral sensory and/or motor neuropathy.
   * Prior treatment with oxaliplatin.
   * Limitation of the patient's ability to comply with the treatment or follow-up protocol.
   * Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
2. Symptomatic, progressive or corticosteroids-requiring documented brain metastases or leptomeningeal disease involvement.
3. Men or women of childbearing potential who are not using an effective method of contraception as previously described; women who are pregnant or breast feeding.
4. Patients who have had RT in more than 35% of the bone marrow.
5. Treatment with any investigational product within 30 days before the first infusion.
6. Prior treatment with PM060184.
7. Prior treatment with gemcitabine-containing therapy for advanced disease (adjuvant therapy is allowed, provided not more than six cycles were administered and relapse occurred more than six months after the last drug administration), and/or:

   * Patients who have previously discontinued gemcitabine-containing regimens due to gemcitabine-related toxicity.
8. Known hypersensitivity to gemcitabine or any component of the formulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- New York, New York, United States
- Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 57 patients were enrolled at three investigational sites, and 55 patients were treated with the GEM/PM060184 combination. Two patients were never treated.
  Patients participated in this trial between 12 December 2014 and 11 July 2019 (last follow-up). The first dose of the first cycle was given on 10 February 2015 and the last dose of the last cycle was given on 7 June 2019.
Groups:
- GEM/PM060184 Dose Level I: Patients were to receive GEM first, followed by PM060184, both on Day 1 and Day 8 q3wk.
  Administration of study treatment was as follows:
  * GEM: i.v. infusion over 30 min (± 10 min) via a central or peripheral venous catheter through a pump device, followed by:
  * PM060184: i.v. infusion over 10 min (± 3 min) via a central or peripheral venous catheter through a pump device.
  Dose Level I: 800 mg/m^2 GEM / 6.0 mg/m^2 PM060184
- GEM/PM060184 Dose Level II: Patients were to receive GEM first, followed by PM060184, both on Day 1 and Day 8 q3wk.
  Administration of study treatment was as follows:
  * GEM: i.v. infusion over 30 min (± 10 min) via a central or peripheral venous catheter through a pump device, followed by:
  * PM060184: i.v. infusion over 10 min (± 3 min) via a central or peripheral venous catheter through a pump device.
  Dose Level II: 800 mg/m^2 GEM / 7.0 mg/m^2 PM060184
- GEM/PM060184 Dose Level III: Patients were to receive GEM first, followed by PM060184, both on Day 1 and Day 8 q3wk.
  Administration of study treatment was as follows:
  * GEM: i.v. infusion over 30 min (± 10 min) via a central or peripheral venous catheter through a pump device, followed by:
  * PM060184: i.v. infusion over 10 min (± 3 min) via a central or peripheral venous catheter through a pump device.
  Dose Level III: 1000 mg/m^2 GEM / 6.0 mg/m^2 PM060184
- GEM/PM060184 Dose Level IV: Patients were to receive GEM first, followed by PM060184, both on Day 1 and Day 8 q3wk.
  Administration of study treatment was as follows:
  * GEM: i.v. infusion over 30 min (± 10 min) via a central or peripheral venous catheter through a pump device, followed by:
  * PM060184: i.v. infusion over 10 min (± 3 min) via a central or peripheral venous catheter through a pump device.
  Dose Level IV: 1000 mg/m^2 GEM / 8.0 mg/m^2 PM060184
- GEM/PM060184 Dose Level V: Patients were to receive GEM first, followed by PM060184, both on Day 1 and Day 8 q3wk.
  Administration of study treatment was as follows:
  * GEM: i.v. infusion over 30 min (± 10 min) via a central or peripheral venous catheter through a pump device, followed by:
  * PM060184: i.v. infusion over 10 min (± 3 min) via a central or peripheral venous catheter through a pump device.
  Dose Level V: 1000 mg/m^2 GEM / 9.0 mg/m^2 PM060184
- GEM/PM060184 Dose Level VI: Patients were to receive GEM first, followed by PM060184, both on Day 1 and Day 8 q3wk.
  Administration of study treatment was as follows:
  * GEM: i.v. infusion over 30 min (± 10 min) via a central or peripheral venous catheter through a pump device, followed by:
  * PM060184: i.v. infusion over 10 min (± 3 min) via a central or peripheral venous catheter through a pump device.
  Dose Level VI: 1000 mg/m^2 GEM / 9.3 mg/m^2 PM060184
- GEM/PM060184 Dose Level VII: Patients were to receive GEM first, followed by PM060184, both on Day 1 and Day 8 q3wk.
  Administration of study treatment was as follows:
  * GEM: i.v. infusion over 30 min (± 10 min) via a central or peripheral venous catheter through a pump device, followed by:
  * PM060184: i.v. infusion over 10 min (± 3 min) via a central or peripheral venous catheter through a pump device.
  Dose Level VII:1000 mg/m^2 GEM / 10.0 mg/m^2 PM060184
- GEM/PM060184 Dose Level VIII: Patients were to receive GEM first, followed by PM060184, both on Day 1 and Day 8 q3wk.
  Administration of study treatment was as follows:
  * GEM: i.v. infusion over 30 min (± 10 min) via a central or peripheral venous catheter through a pump device, followed by:
  * PM060184: i.v. infusion over 10 min (± 3 min) via a central or peripheral venous catheter through a pump device.
  Dose Level VIII:1000 mg/m^2 GEM / 10.5 mg/m^2 PM060184
Period: Dose Level I
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Started | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Never Treated | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level II
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Started | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment-related AE | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-treatment-related AE | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Level III
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Started | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Treatment-related AE | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Dose Level IV
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Started | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Period: Dose Level V
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Started | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Period: Dose Level VI
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Started | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 9 | 0 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 7 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Treatment-related AE | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Period: Dose Level VII
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Started | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 16 | 0
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Treatment-related AE | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Period: Dose Level VIII
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Progressive disease | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Treatment-related AE | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Never treated | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII | Total
Number analyzed (Participants) | 5 | 7 | 4 | 5 | 5 | 9 | 16 | 6 | 57
Age, Continuous [Median (Full Range); unit: years] | 56.0 [25 to 69] | 67.0 [54 to 74] | 58.5 [51 to 72] | 65.0 [62 to 68] | 68.0 [44 to 76] | 62.0 [38 to 76] | 59.0 [29 to 80] | 49.0 [33 to 63] | 62.0 [25 to 80]
Age, Customized [Count of Participants; unit: Participants]
  18-55 | 2 | 2 | 2 | 0 | 1 | 3 | 4 | 5 | 19
  56-75 | 3 | 5 | 2 | 5 | 3 | 5 | 11 | 1 | 35
  >75 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 4 | 2 | 5 | 4 | 6 | 15 | 5 | 42
  Male | 4 | 3 | 2 | 0 | 1 | 3 | 1 | 1 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 4 | 1 | 2 | 3 | 5 | 5 | 2 | 26
  Black or African American | 0 | 2 | 0 | 0 | 2 | 2 | 5 | 1 | 12
  Asian | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hispanic/Latino | 0 | 1 | 3 | 3 | 0 | 2 | 5 | 2 | 16
  Not provided/not available | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 3 | 4 | 3 | 5 | 12 | 4 | 36
  Spain | 4 | 3 | 1 | 1 | 2 | 4 | 4 | 2 | 21
ECOG PS [Count of Participants; unit: Participants] — ECOG PS, Eastern Cooperative Oncology Group performance status PS 0 Fully active able to carry on all pre-disease performance without restriction PS 1 Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature PS 2 Ambulatory and capable of all selfcare but unable to carry out any work activities up and about more than 50% of waking hours PS 3 Capable of only limited selfcare confined to bed or chair more than 50% of waking hours PS 4 Completely disabled cannot carry on any selfcare; totally confined to bed or chair PS 5 Dead
  Participants
    0 | 1 | 1 | 0 | 0 | 3 | 2 | 5 | 3 | 15
    1 | 4 | 6 | 4 | 5 | 2 | 7 | 11 | 3 | 42
Body surface area [Median (Full Range); unit: m^2] | 1.6 [1.4 to 2.0] | 1.7 [1.5 to 1.9] | 2.0 [1.7 to 2.0] | 1.7 [1.5 to 1.9] | 1.9 [1.8 to 2.1] | 1.8 [1.4 to 2.1] | 1.8 [1.4 to 2.1] | 1.6 [1.5 to 2.2] | 1.8 [1.4 to 2.2]
Tumor type [Count of Participants; unit: Participants]
  NSCLC | 3 | 5 | 1 | 2 | 1 | 3 | 3 | 0 | 18
  Gynecological (endometrial or cervical) | 0 | 2 | 0 | 1 | 0 | 3 | 6 | 1 | 13
  Epithelial ovarian cancer | 0 | 0 | 2 | 1 | 3 | 1 | 5 | 1 | 13
  Breast cancer | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 4
  GIST | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 3
  Head and neck cancer | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 3
  GCTs | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Adenocarcinoma or carcinoma of unknown primary site | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Time from diagnosis to first infusion [Median (Full Range); unit: months] | 30.2 [10.9 to 58.4] | 43.0 [7.3 to 76.3] | 23.2 [9.2 to 59.4] | 34.3 [6.2 to 88.6] | 23.4 [14.3 to 111.3] | 33.9 [12.0 to 178.1] | 44.5 [14.0 to 110.0] | 48.8 [14.0 to 110.0] | 48.8 [25.2 to 207.1]
Time from last progressive disease to first infusion [Median (Full Range); unit: months] | 1.6 [0.9 to 2.0] | 1.0 [0.3 to 2.2] | 2.2 [1.2 to 3.5] | 1.7 [0.5 to 2.2] | 1.4 [0.1 to 2.2] | 2.4 [0.1 to 3.5] | 1.2 [0.6 to 9.3] | 0.7 [0.0 to 2.5] | 1.4 [0.0 to 9.3]
Time-to-progression of last prior therapy [Median (Full Range); unit: months] | 1.6 [0.9 to 18.4] | 3.8 [1.4 to 18.2] | 3.4 [1.4 to 4.9] | 6.7 [1.8 to 9.7] | 11.7 [2.3 to 13.6] | 5.4 [1.6 to 48.1] | 3.0 [1.6 to 22.3] | 2.9 [1.7 to 4.6] | 3.7 [0.9 to 48.1]
Bulky disease [Count of Participants; unit: Participants] — Bulky disease is defined as any target lesion measuring at least 50 mm
  Participants | 1 | 1 | 1 | 0 | 1 | 3 | 5 | 2 | 14
Site involvement at baseline [Median (Full Range); unit: sites] | 3 [2 to 5] | 4 [2 to 5] | 4.5 [3 to 5] | 3 [2 to 6] | 3 [1 to 5] | 4 [2 to 7] | 4 [1 to 7] | 3.5 [2 to 4] | 4 [1 to 7]
Lines of prior anticancer therapies [Median (Full Range); unit: lines] | 2 [1 to 5] | 3 [1 to 6] | 3 [2 to 5] | 2 [1 to 6] | 3 [1 to 6] | 3 [2 to 3] | 3 [2 to 7] | 3.5 [2 to 6] | 3 [1 to 7]
Agents of prior anticancer therapies [Median (Full Range); unit: Agents] | 4 [2 to 6] | 4 [2 to 7] | 4.5 [4 to 6] | 5 [3 to 8] | 3 [3 to 8] | 3 [2 to 6] | 4.5 [3 to 8] | 5 [3 to 9] | 4 [2 to 9]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities
Description: Dose-limiting toxicities were defined as:
  * Grade 4 neutropenia lasting >3 days
  * Grade≥3 febrile neutropenia of any duration or neutropenic sepsis
  * Grade 4 thrombocytopenia or grade 3 with any major bleeding episode requiring a platelet transfusion
  * Grade 4 ALT/AST increase, or grade 3 lasting >7 days
  * Treatment-related grade≥2 ALT/AST increase concomitantly with ≥2 x ULN total bilirubin increase and normal AP
  * Any other grade≥3 non-hematological AE that was suspected to be related to study drugs, except nausea/vomiting, hypersensitivity reactions, extravasations, grade 3 asthenia lasting less than one week, anorexia, and non-clinically relevant isolated biochemical abnormalities
  * Delay in the administration of Cycle 2 of the combination exceeding seven (+1) days of the treatment due date due to any AEs related to study drugs.
  * The following circumstances were to be discussed between the Principal Investigator and the Sponsor, and the final consensus had to be documented
Time Frame: From the start of treatment to the end of cycle one which are 3 weeks
Population: Thirteen patients were not evaluable: 11 patients because they did not complete Cycle 1, and two patients because they were withdrawn from the study before receiving the first study drug infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Number analyzed (Participants) | 3 | 6 | 3 | 3 | 4 | 7 | 13 | 5
Participants | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1

2. Secondary Outcome: Number of Participants With Clinical Benefit
Description: Clinical benefit defined as any response or stable disease ≥4 months. Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression). Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Every two cycles (every six weeks ± one week) until Cycle 4, and then every three cycles (every nine weeks ± one week) while on treatment, up to 2 years
Population: Eleven patients were not evaluable: nine patients because they were withdrawn from the study before undergoing a tumor assessment, and two patients because they were withdrawn from the study before receiving the first study drug infusion
Measure: Count of Participants; unit: Participants
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
Number analyzed (Participants) | 4 | 6 | 3 | 4 | 4 | 9 | 11 | 5
Participants | 1 | 3 | 2 | 1 | 1 | 2 | 6 | 2

ADVERSE EVENTS:
Time Frame: Participants were assessed through study completion, approximately 2 years
Description: Two patients were never treated with plitidepsin and were excluded from the analysis of safety.
Arm/Group | GEM/PM060184 Dose Level I | GEM/PM060184 Dose Level II | GEM/PM060184 Dose Level III | GEM/PM060184 Dose Level IV | GEM/PM060184 Dose Level V | GEM/PM060184 Dose Level VI | GEM/PM060184 Dose Level VII | GEM/PM060184 Dose Level VIII
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/7 | 0/4 | 0/5 | 1/5 | 0/9 | 5/16 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/4 | 3/7 | 2/4 | 1/5 | 3/5 | 3/9 | 8/16 | 4/5
Other Adverse Events (participants affected / at risk) | 4/4 | 7/7 | 4/4 | 5/5 | 5/5 | 9/9 | 16/16 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEM/PM060184 Dose Level I (N=4) | GEM/PM060184 Dose Level II (N=7) | GEM/PM060184 Dose Level III (N=4) | GEM/PM060184 Dose Level IV (N=5) | GEM/PM060184 Dose Level V (N=5) | GEM/PM060184 Dose Level VI (N=9) | GEM/PM060184 Dose Level VII (N=16) | GEM/PM060184 Dose Level VIII (N=5)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GEM/PM060184 Dose Level I (N=4) | GEM/PM060184 Dose Level II (N=7) | GEM/PM060184 Dose Level III (N=4) | GEM/PM060184 Dose Level IV (N=5) | GEM/PM060184 Dose Level V (N=5) | GEM/PM060184 Dose Level VI (N=9) | GEM/PM060184 Dose Level VII (N=16) | GEM/PM060184 Dose Level VIII (N=5)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subclavian vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 1 (1) | 1 (1) | 1 (5) | 1 (2) | 2 (7) | 4 (9) | 3 (5) | 1 (2)
Fatigue (General disorders) | 1 (1) | 5 (11) | 3 (8) | 3 (6) | 3 (12) | 2 (4) | 10 (27) | 3 (8)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 2 (3) | 2 (4) | 1 (1)
Mucosal inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (4) | 1 (1)
Catheter site erythema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Feeling of body temperature change (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infusion site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 2 (2) | 0 (0) | 2 (4) | 1 (1) | 1 (1) | 8 (10) | 2 (3)
Breath sounds abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Creatinine renal clearance decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 2 (4) | 2 (3) | 1 (1) | 1 (1) | 3 (14) | 7 (28) | 3 (6)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 2 (7)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 2 (6) | 0 (0)
Lymph node pain (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3) | 2 (3) | 2 (2) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 1 (2) | 1 (12) | 0 (0) | 1 (3) | 1 (3) | 2 (3) | 0 (0)
Neurotoxicity (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 0 (0)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 6 (9) | 2 (4)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 6 (9) | 2 (6)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 2 (2) | 4 (5) | 8 (13) | 4 (9)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (4) | 1 (2) | 2 (2) | 1 (1) | 2 (5) | 8 (20) | 2 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (7) | 5 (7) | 0 (0) | 2 (2) | 4 (8) | 4 (5) | 11 (17) | 4 (8)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (4) | 1 (2) | 1 (1) | 2 (2) | 2 (4) | 6 (9) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 3 (5) | 1 (1)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth loss (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urethritis noninfective (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (3) | 1 (1) | 2 (2) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 3 (4) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (4) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 2 (2) | 2 (2) | 11 (21) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Conjunctivitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is more than 60 days but less than or equal to 180 days from the time submitted to the sponsor for review.

DOCUMENTS (2):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT02533674/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-23): https://cdn.clinicaltrials.gov/large-docs/74/NCT02533674/SAP_001.pdf